CLINICAL TRIAL: NCT00524043
Title: A Randomized, Double-Blind, Placebo- and Active-Controlled, Parallel-Group Study to Evaluate the Efficacy and Safety of a Fixed Dosage of 1.5 mg/Day of Paliperidone Extended Release (ER) in the Treatment of Subjects With Schizophrenia
Brief Title: An Efficacy and Safety Study of One Dosage of Paliperidone Extended Release (ER) in Treating Patients With Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR013771; R076477SCH4012
Record Dates: First submitted 2007-08-30; First posted 2007-09-03 (Estimated); Results first posted 2010-02-26 (Estimated); Last update posted 2014-06-04 (Estimated); Status verified 2014-05

CONDITIONS: Schizophrenia
Keywords: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Paliperidone Palmitate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- 001 (Experimental): Paliperidone ER 1.5 mg tablet once daily for 6 weeks
  Interventions: Drug: Paliperidone ER
- 002 (Active Comparator): Paliperidone ER 6 mg tablet once daily for 6 weeks
  Interventions: Drug: Paliperidone ER
- 003 (Placebo Comparator): Placebo Once daily for 6 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Paliperidone ER — 1.5 mg tablet once daily for 6 weeks
  Arms: 001
Drug: Placebo — Once daily for 6 weeks
  Arms: 003
Drug: Paliperidone ER — 6 mg tablet once daily for 6 weeks
  Arms: 002

SUMMARY:
The purpose of this study is to assess the efficacy and safety of 1.5 mg/day dose of paliperidone Extended Release (ER) as compared with placebo when used to treat patients with schizophrenia.

DETAILED DESCRIPTION:
Currently, treatment of acute symptoms in schizophrenia is less than ideal, up to one-third of patients with schizophrenia do not respond to current treatments, and poor drug tolerability can decrease a patient's ability to remain on treatment. Paliperidone ER doses in the range of 3 mg/day to 12 mg/day have been approved for the treatment of patients with schizophrenia. A lower dosage form of paliperidone ER be efficacious and may reduce the risk of certain adverse effects. This study will evaluate the efficacy of 1 fixed (ie, it does not change during the study) dosage of paliperidone ER (1.5 mg/day) compared with placebo. One fixed dosage of paliperidone ER (6.0 mg/day) will be given to some patients as an active (it has already been shown to have efficacy) control. This is a multicenter, double-blind (neither the patient nor the study-site personnel know which treatment the patient is receiving), randomized (patients are assigned to a treatment group by chance), placebo-controlled (some patients will receive placebo and no active drug), parallel-group (patients in all groups follow the same study design) study in adults who were diagnosed with schizophrenia at least 1 year before screening and who are experiencing an acute episode. The study starts with an up-to-5-day screening phase to find out if the patient is eligible for the study. The screening phase includes a 3- to 5-day washout (the medication dosage is tapered down and finally stopped) of any medications that are being taken by a patient but that are not allowed during the study. A 6-week double-blind treatment phase follows and finishes with an end-of-study visit. A post-study visit to collect additional safety data will be scheduled for 1 week after a patient receives his or her last dose of study drug. The length of the entire study is about 8 weeks. Patients who withdraw from the study before completing the double-blind treatment phase will complete the end-of-study visit procedures at the time they withdraw and the post-study visit 1 week after receiving their last dose of study drug. For all patients leaving the study, the investigator will make every effort to see that they receive adequate continuity of care. At baseline (the visit just before a patient takes the first dose of study drug), all patients will be randomly assigned to 1 of the 3 possible treatment groups to receive paliperidone ER 1.5 mg/day, paliperidone ER 6 mg/day, or placebo once daily for 6 weeks. Patients must be voluntary inpatients at the time of randomization, and they must remain in the hospital for a minimum of 8 days. Efficacy will be measured using the following rating scales: the Positive and Negative Syndrome Scale (PANSS), the Clinical Global Impression-Severity (CGI-S), the Personal and Social Performance Scale (PSP), and the Medical Outcomes Study Short Form Health Survey-36 (MOS SF-36). Safety will be evaluated using physical examinations, ECGs, clinical laboratory testing (hematology, serum chemistry, and urinalysis), testings for pregnancy, and monitoring for adverse events including extrapyramidal symptoms (EPS) using the Abnormal Involuntary Movement Scale (AIMS), Barnes Akathisia Rating Scale (BARS), and Simpson-Angus Rating Scale (SAS). The study hypothesis is that Paliperidone ER at 1.5 mg per day will be effective in the treatment of schizophrenia as measured by the change in total PANSS score between baseline and endpoint in comparison with placebo. Oral paliperidone ER 1.5 mg or 6.0 mg tablets or matching oral placebo tablets taken once daily in the morning for 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with schizophrenia according to the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) (295.10, 295.20, 295.30, 295.60, 295.90) at least 1 year before screening
* Experiencing an acute episode with a total PANSS score at screening of between 70 and 120
* Are otherwise physically healthy
* Agree to at least 8 days of voluntary hospitalization.

Exclusion Criteria:

* Active comorbid DSM-IV axis I diagnosis other than schizophrenia (nicotine and caffeine dependence are not exclusionary)
* Treatment with antidepressants (unless a subject has been on a stable dosage for at least 3 months before baseline) other than monoamine oxidase inhibitors
* DSM-IV diagnosis of substance dependence within 6 months before screening evaluation (nicotine and caffeine dependence are not exclusionary)
* Any medical condition that could potentially alter the absorption, metabolism, or excretion of the study medication, such as Crohn's disease, liver disease, or renal disease
* Relevant history of any significant or unstable cardiovascular, respiratory, neurologic (including seizures or significant cerebrovascular), renal, hepatic, endocrine, or immunologic disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2007-09; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (20):
- United States (12):
  - Cerritos, California
  - Torrance, California
  - Washington D.C., District of Columbia
  - Bradenton, Florida
  - Leesburg, Florida
  - Atlanta, Georgia
  - Rockville, Maryland
  - Nutley, New Jersey
  - Cedarhurst, New York
  - Hollis, New York
  - Moore, Oklahoma
  - Austin, Texas
- India (5):
  - Calicut
  - Hyderabad
  - Mumbai
  - Pune
  - Varanasi
- Taiwan (3):
  - Hualien City
  - Tainan
  - Taipei

REFERENCES:
- See also: A Study of the Efficacy and Safety of One Dosage of Paliperidone Extended Release (ER) in Treating Patients With Schizophrenia — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=72&filename=CR013771_CSR.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study began on 21 September 2007 when the first patient was enrolled and ended on 20 November 2008 when the last patient left the study. The study was performed at medical clinics in the United States, India, and Taiwan.
Pre-assignment Details: Patients who wished to enter the study were screened and, if necessary, had prohibited medications (such as other antipsychotic drugs) washed out for 3 to 5 days before beginning the study. Eligible patients were excluded prior to beginning the study if, for example, they took a prohibited medication.
Groups:
- Placebo: One oral placebo tablet daily for 6 weeks.
- Paliperidone ER 6 mg: Active comparator. One 6 mg oral tablet daily for 6 weeks. The 6 mg dose of paliperidone ER has been shown to have efficacy in previous studies.
- Paliperidone ER 1.5 mg: Experimental dose of paliperidone ER. One 1.5 mg oral tablet daily for 6 weeks.
Period: Overall Study
Arm/Group | Placebo | Paliperidone ER 6 mg | Paliperidone ER 1.5 mg
Started | 64 (One patient was randomly assigned to treatment but did not receive placebo.) | 70 | 66
Completed | 34 | 42 | 35
Not Completed | 30 | 28 | 31
Not completed — Lack of Efficacy | 15 | 13 | 14
Not completed — Withdrawal by Subject | 5 | 7 | 7
Not completed — Adverse Event | 5 | 2 | 7
Not completed — Lost to Follow-up | 3 | 5 | 3
Not completed — Various (eg, incarceration) | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Paliperidone ER 6 mg | Paliperidone ER 1.5 mg | Total
Number analyzed (Participants) | 64 | 70 | 66 | 200
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 64 | 70 | 66 | 200
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.5 (11.57) | 40.3 (12.84) | 41.3 (10.96) | 39.4 (11.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 23 | 16 | 57
  Male | 46 | 47 | 50 | 143
Region of Enrollment [Number; unit: participants]
  India | 23 | 25 | 24 | 72
  Taiwan | 7 | 12 | 9 | 28
  United States | 34 | 33 | 33 | 100

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in PANSS Total Score at the End of the Double-blind Treatment Phase (Week 6 or the Last Assessment Obtained After the Baseline Assessment).
Description: The Positive and Negative Syndrome Scale (PANSS) is a tool used by psychiatrists to measure the symptoms of psychosis experienced by a patient with schizophrenia. It includes 30 items that produce a total score ranging from a minimum of 30 (indicating least severe symptoms of illness) to a maximum of 120 (indicating most severe symptoms of illness). A negative change in score from baseline to end point indicates improvement in the symptoms of illness.
Time Frame: Baseline, 6 weeks
Population: The intent-to-treat analysis set included all enrolled patients who received at least 1 dose of paliperidone ER or placebo and had both the baseline and at least 1 postbaseline efficacy assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Paliperidone ER 6 mg | Paliperidone ER 1.5 mg
Number analyzed (Participants) | 63 | 70 | 66
units on a scale | -11.7 (22.84) | -15.0 (26.02) | -8.9 (25.41)
Statistical Analysis 1: Comparison: Placebo vs Paliperidone ER 1.5 mg; Sample size estimation was based on the assumption that the difference between the paliperidone ER 1.5 mg dose group and the placebo group in the mean change in PANSS total score from baseline to end point was 11 points with a within-group standard deviation of 20 points. It was calculated that 65 patients were needed per treatment group to detect a statistically significant treatment difference between the paliperidone ER 1.5 mg dose group and the placebo group with a power of 87.5%; Test type: Superiority or Other; p = 0.504, ANCOVA — Based on ANCOVA model with treatment (Placebo, Paliperidone ER 1.5 mg, and Paliperidone ER 6 mg) and country as factors, and baseline value as a covariate. Comparison with placebo was without multiplicity adjustment; Mean Difference (Final Values) = 2.8, 95% CI [-5.47 to 11.09], Standard Error of Mean 4.20
Statistical Analysis 2: Comparison: Placebo vs Paliperidone ER 6 mg; Test type: Superiority or Other; p = 0.431, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Paliperidone ER 6 mg was used for assay sensitivity; Mean Difference (Final Values) = -3.3, 95% CI [-11.46 to 4.90], Standard Error of Mean 4.15

2. Secondary Outcome: Change From Baseline to the End of the Double-blind Treatment Phase (Week 6 or the Last Assessment Obtained After the Baseline Assessment) in CGI-S
Description: The Clinical Global Impression-Severity (CGI-S) rating scale is used by psychiatrists to rate the severity of a patient's psychotic condition on a 7-point scale ranging from 1 (not ill) to 7 (extremely severe). The scale permits a global evaluation of the patient's condition at a given time.
Time Frame: Baseline, 6 weeks
Population: as for outcome 1
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Placebo | Paliperidone ER 6 mg | Paliperidone ER 1.5 mg
Number analyzed (Participants) | 63 | 70 | 66
units on a scale | -1.0 [-2 to 2] | -0.5 [-3 to 2] | 0.0 [-3 to 2]
Statistical Analysis 1: Comparison: Placebo vs Paliperidone ER 1.5 mg; Test type: Superiority or Other; p = 0.626, ANCOVA — Based on ANCOVA model on ranks with treatment (Placebo, Paliperidone ER 1.5 mg, and Paliperidone ER 6 mg) and country as factors, and baseline value as a covariate. Comparison with placebo was without multiplicity adjustment

3. Secondary Outcome: Change From Baseline to End Point (Week 6 or the Last Assessment After the Baseline Assessment) in PSP Score
Description: The Personal and Social Performance (PSP) scale assesses the degree of difficulty (ranging from i [absent] to vi [very severe]) a patient exhibits over a 1-month period in socially useful activities, personal and social relationships, self care, and disturbing and aggressive behavior. The overall score ranges from 1 to 100. Patients with scores of 71 to 100 have a mild degree of difficulty; patients with scores from 31 to 70 have various degrees of disability; and patients with scores of 30 or less function so poorly as to require intensive supervision.
Time Frame: Baseline, 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Paliperidone ER 6 mg | Paliperidone ER 1.5 mg
Number analyzed (Participants) | 63 | 70 | 66
units on a scale | 1.6 (17.09) | 5.7 (13.39) | 2.9 (14.37)
Statistical Analysis 1: Comparison: Placebo vs Paliperidone ER 1.5 mg; Test type: Superiority or Other; p = 0.870, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.4, 95% CI [-4.86 to 5.74], Standard Error of Mean 2.69

4. Secondary Outcome: Change From Baseline to End Point (Week 6 or the Last Assessment After the Baseline Assessment) in MOS SF-36 Physical Component Summary Scale Score
Description: The Medical Outcomes Study Short Form Health Survey-36 (MOS SF-36) is a measure of patient-reported health status. It is a 36-item questionnaire measuring 8 domains (physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health). Each domain score ranges from 0 (worst) to 100 (best), with higher scores reflecting better health-related functional status. Two summary scale scores are computed based on weighted combinations of the 8 subscale scores: the Physical Component Summary and the Mental Component Summary.
Time Frame: Baseline, 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Paliperidone ER 6 mg | Paliperidone ER 1.5 mg
Number analyzed (Participants) | 63 | 70 | 66
units on a scale | 0.4 (6.94) | 0.6 (9.45) | -0.2 (9.79)
Statistical Analysis 1: Comparison: Placebo vs Paliperidone ER 1.5 mg; Test type: Superiority or Other; p = 0.126, ANCOVA — Based on ANCOVA model with treatment (placebo, paliperidone ER 1.5 mg, and paliperidone ER 6 mg) and country as factors and baseline value as a covariate. Comparison with placebo was without multiplicity adjustment

5. Secondary Outcome: Change From Baseline to End Point (Week 6 or the Last Assessment After the Baseline Assessment) in MOS SF-36 Mental Component Summary Scale Score
Description: The MOS SF-36 is a measure of patient-reported health status. It is a 36-item questionnaire measuring 8 domains (physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health). Each domain score ranges from 0 (worst) to 100 (best), with higher scores reflecting better health-related functional status. Two summary scale scores are computed based on weighted combinations of the 8 domain scores: the Physical Component Summary and the Mental Component Summary.
Time Frame: Baseline, 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Paliperidone ER 6 mg | Paliperidone ER 1.5 mg
Number analyzed (Participants) | 63 | 70 | 66
units on a scale | 3.5 (13.14) | 6.1 (13.39) | 2.1 (11.71)
Statistical Analysis 1: Comparison: Placebo vs Paliperidone ER 1.5 mg; Test type: Superiority or Other; p = 0.691, ANCOVA — [p-value comment as in outcome 4, analysis 1]

ADVERSE EVENTS:
Time Frame: Up to 8 weeks, including the screening period (2 to 6 days), the 6-week treatment period, and 1 week follow up. Monitoring for adverse events began after the patient was enrolled and continued until the last study-related procedure was performed.
Description: There were 65 patients randomly assigned to treatment with placebo, but 1 patient in the Placebo group did not receive any treatment. Thus any adverse events experienced by this subject are not reported here.
Arm/Group | Placebo | Paliperidone ER 6 mg | Paliperidone ER 1.5 mg
Serious Adverse Events (participants affected / at risk) | 7/64 | 5/70 | 7/66
Other Adverse Events (participants affected / at risk) | 21/64 | 29/70 | 19/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=64) | Paliperidone ER 6 mg (N=70) | Paliperidone ER 1.5 mg (N=66)
Psychotic disorder (Psychiatric disorders) | 6 (6) | 2 (2) | 4 (4)
Schizophrenia (Psychiatric disorders) | 0 (0) | 2 (2) | 2 (2)
Aggression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=64) | Paliperidone ER 6 mg (N=70) | Paliperidone ER 1.5 mg (N=66)
Insomnia (Psychiatric disorders) | 6 (11) | 7 (10) | 9 (11)
Headache (Nervous system disorders) | 10 (11) | 8 (11) | 5 (7)
Tremor (Nervous system disorders) | 2 (2) | 7 (7) | 2 (2)
Dizziness (Nervous system disorders) | 1 (2) | 2 (2) | 5 (5)
Akathisia (Nervous system disorders) | 1 (1) | 4 (4) | 0 (0)
Constipation (Gastrointestinal disorders) | 4 (5) | 6 (9) | 3 (3)
Vomiting (Gastrointestinal disorders) | 0 (0) | 4 (5) | 1 (2)

LIMITATIONS AND CAVEATS:
No information from this study about efficacy and safety with treatment beyond 6 weeks. Study not designed to establish efficacy of 6 mg dose relative to 1.5 mg dose. No information on efficacy of paliperidone ER doses between 1.5 and 3 mg.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days